CLINICAL TRIAL: NCT04436692
Title: Dietary Intervention in Overweight Subjects With Intellectual Disabilties Using the Nudging Approach as Method
Brief Title: Dietary Intervention and Adults With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Svein Olav Kolset, Professor, University of Oslo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Department of Nutrition
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-05

CONDITIONS: Intellectual Disabilities Nutritional; Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Improve dietary pattern (Other): Nudging approach to test this methodological approach in persons with intellectual disabilitites with goal to improve dietary pattern and loss of weight
  Interventions: Behavioral: Nudging

INTERVENTIONS:
Behavioral: Nudging — Use nudging approach by using smaller plates and glasses and increasing the availability of fruits and vegetables

SUMMARY:
Goal The overall aim of the study is to improve the health of persons with Intellectual disabilities

DETAILED DESCRIPTION:
Purpose

There are two main purposes of the study The first is to study the diet and heath of persons with intellectual disabilities. The second is to increase their knowledge on nutrition and health and that of service providers in municipalities housing facilities and to test, in an intervention, the effects of a method for weight reduction in adult persons with intellectual disabilities with overweight and obesity. Physical activity is also an important factor in weight reduction, but this study focuses only on nutrition, to obtain new information on this one factor in weight reduction. A combined study with many changes in a short period of time is very challenging for the group in question.

The vision is that results from this study will lead to improved health promotive and preventive services in the municipality in the future, to adult persons with intellectual disabilities and that this study also can have effects on services also for other groups, such as those with the fields of psychiatry and drug problems.

ELIGIBILITY:
Inclusion criteria:

* Mild intellectual disability and overweight
* Moderate intellectual disability and overweight

Exclusion Criteria:

* Metabolic diseases
* Hypertension
* Diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in body weight by using a nudging approach in adults with intellectual disabilities | One year
  2 kg weight decrease

SECONDARY OUTCOMES:
Change in consumption of fruits and vegetables as measured using dietary survey | One year
  Dietary change 1

OTHER OUTCOMES:
Change in consumption of sugar containing beverages as measured using dietary survey | One year
  Dietary change 2

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Andersen, PhD, Study Chair — Institute of Basic Medical Sciences
Locations (1):
- University of Oslo, Oslo, Norway